CLINICAL TRIAL: NCT01972282
Title: Registry on WATCHMAN Outcomes in Real-Life Utilization
Acronym: EWOLUTION
Status: Completed | Type: Observational
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: EWOLUTION; 90875647 (Other: Boston Scientific)
Record Dates: First submitted 2013-10-24; First posted 2013-10-30 (Estimated); Results first posted 2019-05-07 (Actual); Last update posted 2019-05-07 (Actual); Status verified 2018-05

CONDITIONS: Patients With Atrial Fibrillation at Risk for Thrombus Formation, Thromboembolism, Stroke
Keywords: Atrial fibrillation; Stroke; Thrombus; Thromboembolism; Left atrial appendage
MeSH Terms: conditions — Thromboembolism; Stroke; Atrial Fibrillation; Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: WATCHMAN Left Atrial Appendage Closure

SUMMARY:
The WATCHMAN LAA Closure Technology is designed to prevent embolization of thrombi that may form in the LAA, thereby preventing the occurrence of ischemic stroke and systemic thromboembolism. The objectives of this observational, prospective, non-randomized multicenter study are (1) to compile real-world clinical outcomes data for WATCHMAN LAA (left atrial appendage) Close Technology in patients who are implanted with the WATCHMAN device in a commercial clinical setting and (2) to collect real-world usage data that may be needed for reimbursement of WATCHMAN technology in certain countries.

DETAILED DESCRIPTION:
Approximately 1000 subjects will be enrolled in the study. To reduce the impact of individual center bias, each site may include up to 45 subjects and each country may include a maximum of 500 patients. Up to 70 sites (international, outside of US) will participate in the study.

Primary analyses may include, but will not be limited to, the following: procedural complications, incidence of stroke and death. Descriptive statistics will be used for baseline, procedure and follow-up data collected through the study.

Each patient will be followed for a period of two years after enrollment according to the schedule and standard practice at the enrolling centers. There will be no additional visits, nor procedures, for subjects who participate in the study. Subjects are expected to be followed at implant, then at one post-implant visit (typically between 1-3 months of implant), and then annually through 2 years post implant. An intermediate visit may be scheduled in a number of patients, per physician discretion. In order to reliably capture patient status at study end, a follow-up window of 24 +/- 3 months will be considered acceptable for scheduling the last visit.

For subjects who are not scheduled to visit the clinic for a follow-up, a subject contact (e.g. phone call) will ensure capture of the endpoint related information; however, it is recommended to perform an in-office visit for at least the first annual visit.

Enrollment is expected to be completed in 21 months; therefore, the total study duration is estimated to be 48 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are eligible for a WATCHMAN device according to current international and local guidelines (and future revisions) and per physician discretion;
* Patient who are willing and capable of providing informed consent, participating in all testing associated with this clinical investigation at an approved clinical investigational center;
* Patients whose age is 18 years or above, or of legal age to give informed consent specific to state and national law.

Exclusion Criteria:

* Patient who are currently enrolled in another investigational study or registry that would directly interfere with the current study, except when the patient is participating in a mandatory governmental registry, or a purely observational registry with no associated treatments. Each instance should be brought to the attention of the sponsor to determine eligibility;
* Women of childbearing potential who are, or plan to become, pregnant during the time of the study (method of assessment upon physician's discretion);
* The subject is unable or not willing to complete follow-up visits and examination for the duration of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with non-valvular atrial fibrillation
Sampling Method: Non-Probability Sample
Enrollment: 1025 (Actual)
Dates: Start 2013-10-28 (Actual); Primary Completion 2015-11 (Actual); Study Completion 2018-01-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lucas VA Boersma, Principal Investigator — St. Antonius Hospital
Locations (47):
- OLV Ziekenhuis, Aalst, Belgium
- France (7):
  - Hospitaux du Haut Leveque, Bordeaux
  - CHU Henri Mondor, Créteil
  - University Hospital, Grenoble
  - CHRU Lille, Lille
  - CHU La Timone Hospital, Marseille
  - Nouvelles Cliniques Nantaises, Nantes
  - Groupe hospitalier Bichat Claude Bernard, Paris
- Germany (17):
  - Charite Universitatsmedizin Berlin - Campus Virchow Klinikum - Medizinische Klinik fur Kardiologie, Berlin
  - Vivantes Klinikum Am Urban, Berlin
  - Vivantes Klinikum im Friedrichshain, Berlin
  - Evangelisches Krankenhaus, Bielefeld
  - Universitatklinikum Medizinische, Bonn
  - Dominikus-Krankenhaus, Düsseldorf
  - Elisabeth Krankenhaus, Essen
  - Cardio Vasculares Centrum Sankt Katharinen, Frankfurt
  - Cardioangiologisches Centrum Bethanien, Frankfurt
  - Univeritatsmedizin Greifswald, Greifswald
  - Cardiologicum Hamburg, Hamburg
  - Aklepios Klinik St Georg, Hamburg
  - Universitatklinikum Leipzig, Leipzig
  - Universitatsmedizin Mainz, Mainz
  - Stadtisches Klinikum Neuperlach, Munich
  - Krankenhaus Barmherzige Bruder, Regensburg
  - Asklepios Klinik Weissenfels, Weißenfels
- Beaumont Hospital, Dublin, Ireland
- Italy (4):
  - Ospedale Ferrarotto Alessi, Catania
  - ASL TO 4 Ospedale di Cirie, Cirié
  - Ospedale San Raffaele, Milan
  - Ospedale Sacro Cuore "Don Calabria", Negrar
- Netherlands (4):
  - Medisch Spectrum Twente, Enschede
  - Medisch Centrum Leeuwarden, Leeuwarden
  - St. Antonius Hospital, Nieuwegein
  - Erasmus Medisch Centrum Rotterdam, Rotterdam
- Poland (2):
  - Szpital Uniwersytecki nr 1im dr A Jurasza, Bydgoszcz
  - Clinical Hospital University of Medicine, Poznan
- Hospital de Santa Maria, Lisbon, Portugal
- Russia (3):
  - Regional Vascular Center, Krasnoyarsk
  - State Cardiology Research Center, Moscow
  - State Research Institute of Circulation Pathology, Novosibirsk
- King Fahed Medical City - Prince Salman Cardiac Center, Riyadh, Saudi Arabia
- Hospital Clinico Universitario de Salamanca, Salamanca, Spain
- Al Qassimi Hospital, Sharjah city, United Arab Emirates
- United Kingdom (4):
  - Royal Victoria Hospita, Belfast
  - Royal Brompton & Harefield NHS Trust, London
  - Freeman Hospital, Newcastle
  - John Radcliffe Hospital, Oxford

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Aarnink EW, Ince H, Kische S, Pokushalov E, Schmitz T, Schmidt B, Gori T, Meincke F, Protopopov AV, Betts T, Mazzone P, Grygier M, Sievert H, De Potter T, Vireca E, Stein K, Bergmann MW, Boersma LVA. Incidence and predictors of 2-year mortality following percutaneous left atrial appendage occlusion in the EWOLUTION trial. Europace. 2024 Jul 2;26(7):euae188. doi: 10.1093/europace/euae188. PMID 39082730
- [Derived] Boersma LV, Ince H, Kische S, Pokushalov E, Schmitz T, Schmidt B, Gori T, Meincke F, Protopopov AV, Betts T, Mazzone P, Foley D, Grygier M, Sievert H, De Potter T, Vireca E, Stein K, Bergmann MW; following investigators and institutions participated in the EWOLUTION study. Evaluating Real-World Clinical Outcomes in Atrial Fibrillation Patients Receiving the WATCHMAN Left Atrial Appendage Closure Technology: Final 2-Year Outcome Data of the EWOLUTION Trial Focusing on History of Stroke and Hemorrhage. Circ Arrhythm Electrophysiol. 2019 Apr;12(4):e006841. doi: 10.1161/CIRCEP.118.006841. PMID 30939908

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 1025 patients scheduled for a WATCHMAN implant at 47 centers in 13 countries were enrolled over a time period of 19 months prior to the start of the procedure (Oct 2013 - May 2015)
Pre-assignment Details: 5 patients signed the informed consent but never underwent the implant procedures. Those patients are classified as intents, they are included in epidemiological baseline analyses, but not on the endpoint analysis. 1020 patients underwent the implant procedure and are included in all endpoint analyses, regardless of the success of the implant.
Groups:
- WATCHMAN: Patients who are implanted with the WATCHMAN device in a commercial clinical setting.
Period: Overall Study
Arm/Group | WATCHMAN
Started | 1020
Completed | 1005
Not Completed | 15

BASELINE CHARACTERISTICS:
Population: All enrolled patients are included in Baseline analyses including 5 patients who never underwent the study procedure
Arm/Group | WATCHMAN
Number analyzed (Participants) | 1025
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.4 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 411
  Male | 614
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Russian Federation | 81
  United Kingdom | 58
  United Arab Emirates | 8
  Portugal | 17
  Spain | 20
  Saudi Arabia | 15
  Netherlands | 79
  Belgium | 23
  Ireland | 37
  Poland | 38
  Italy | 56
  France | 61
  Germany | 532
CHADS-VASc [Mean (Standard Deviation); unit: scores on a scale] — Total score used to determine adjusted stroke rate, based on the number of risk factors presented by a patient. The higher the number of risk factors, the higher the risk of stroke. Range of score: 0 (lower risk) - 9 (higher risk).
  CHA2DS2-VASc = Congestive heart failure (1 point), Hypertension (1 point), Age ≥75 years (2 points), Diabetes (1 point), Prior Stroke or TIA or thromboembolism (2 points), Vascular disease (1 point), Age 65-74 years (1 point), Sex category (female) (1 point).
  scores on a scale | 4.5 (1.6)
HAS-BLED [Mean (Standard Deviation); unit: scores on a scale] — Score To Assess 1-Year Risk of Major Bleeding in Patients With Atrial Fibrillation, based on the number of risk factors presented by a patient. The higher the number of risk factors, the higher the risk of major bleeding. Range of score: 0 (lower risk) - 9 (higher risk).
  HAS-BLED = Hypertension, Abnormal Renal function, Abnormal Liver function, Stroke, Bleeding, Labile INR, Elderly: Age >65, Concomitant use of Drugs, Alcohol abuse (1 point each)
  scores on a scale | 2.3 (1.2)

OUTCOME MEASURES:

1. Primary Outcome: Procedural Complications
Description: All device/procedure related Serious Adverse Events (with or without Major intervention)
Time Frame: 7 days post-implant
Measure: Number; unit: percentage of participants
Arm/Group | WATCHMAN
Number analyzed (Participants) | 1020
percentage of participants | 2.8

2. Primary Outcome: Ischemic Stroke
Description: occurence of Ischemic stroke during the 2 years of FU. Expressed as nr events / 100 patient-years of FU
Time Frame: 2 year follow-up
Population: Patients who undergo WATCHMAN implant procedure in a commercial clinical setting
Measure: Number (95% Confidence Interval); unit: Nr events/100 Patient-years
Arm/Group | WATCHMAN
Number analyzed (Participants) | 1020
Nr events/100 Patient-years | 1.26 [0.79 to 1.90]

3. Primary Outcome: Death
Description: All cause mortality
Time Frame: 2 year follow-up
Population: Patients who undergo WATCHMAN implant in a commercial clinical setting.
Measure: Count of Participants; unit: Participants
Arm/Group | WATCHMAN
Number analyzed (Participants) | 1020
Participants | 161

ADVERSE EVENTS:
Time Frame: 2 years
Description: Overall number of participants who died due to any cause
Arm/Group | WATCHMAN
All-Cause Mortality (participants affected / at risk) | 161/1020
Serious Adverse Events (participants affected / at risk) | 26/1020
Other Adverse Events (participants affected / at risk) | 0/1020
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | WATCHMAN (N=1020)
Procedural Device/Procedure related Serious Adverse Events (Cardiac disorders) | 26 (1020) — Bleeding; Hematoma; groin vascular damage; device embolization; incomplete seal at device release; pericardial effusion/tamponade; respiratory insufficiency; coronary air embolism; cerebral air embolism; hypotension; adverse reaction to anaesthesia

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-10-03): https://cdn.clinicaltrials.gov/large-docs/82/NCT01972282/Prot_SAP_000.pdf